CLINICAL TRIAL: NCT05949034
Title: Effects of E-Cigarettes in Menthol Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-19-00325
Record Dates: First submitted 2019-05-29; First posted 2023-07-17 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: E-cigarette Use; Smoking Behaviors
Keywords: menthol; cigarette; smoking
MeSH Terms: conditions — Vaping; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- E-Cigarette Flavor 1 Condition (Experimental): Participants will self-administer a flavored e-cigarette.
  Interventions: Device: JUUL E-Cigarette Device
- E-Cigarette Flavor 2 Condition (Experimental): Participants will self-administer a flavored e-cigarette.
  Interventions: Device: JUUL E-Cigarette Device
- E-Cigarette Flavor 3 Condition (Experimental): Participants will self-administer a flavored e-cigarette.
  Interventions: Device: JUUL E-Cigarette Device

INTERVENTIONS:
Device: JUUL E-Cigarette Device — We will use the commercially available and popular JUUL e-cigarette device and e-cigarette solutions.

SUMMARY:
The current laboratory study examines e-cigarette preferences and smoking behaviors in menthol cigarette smokers.

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette smoking for at least the past 2 years
* Interest in trying e-cigarettes
* Report smoking mentholated cigarettes

Exclusion Criteria:

-- Pregnancy and/or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Preference Ratings | 1 hour
  Self-report measures of product preference will be completed following the e-cigarette self-administration. Scores can range from 0 to 100 for the preference rating, with lower scores representing less preference and higher scores representing higher preference.
Mood - Positive Affect Negative Affect Schedule | 4 hours
  This measure is obtained through the completion of the Positive Affect Negative Affect Schedule. A total score will be calculated for both Positive and Negative Affect. Scores can range from 10 to 50 for both the Positive and Negative Affect, with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Mood - Profile of Mood States | 4 hours
  This measure is obtained through the completion of the Profile of Mood States. A total score will be calculated. Scores can range from 10 to 260, with the lower scores representing lower levels of mood disturbance and higher scores representing higher levels of mood disturbance.
Cigarette Craving | 4 hours
  This measure is obtained through the completion of the Brief Questionnaire of Smoking Urges. A total score will be calculated. Scores can range from 10 to 70, with the lower scores representing a lower level of cigarette craving and higher scores representing greater levels of cigarette craving.
Nicotine Withdrawal - Minnesota Nicotine Withdrawal Scale | 4 hours
  This measure is obtained through the completion of the Minnesota Nicotine Withdrawal Scale. A total score will be calculated. Scores can range from 0 to 32, with the lower scores representing a lower level of nicotine withdrawal and higher scores representing greater levels of nicotine withdrawal.
Nicotine Withdrawal - Wisconsin Smoking Withdrawal Scale | 4 hours
  This measure is obtained through the completion of the Wisconsin Smoking Withdrawal Scale. A total score will be calculated. Scores can range from 0 to 112, with the lower scores representing a lower level of nicotine withdrawal and higher scores representing greater levels of nicotine withdrawal.
Smoking Motivation | 2 hours after experimental session outset
  This measure is obtained through the completion of a computerized behavioral task.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Leventhal, Ph.D., Study Chair — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No